CLINICAL TRIAL: NCT03025347
Title: Effect of Exercise on Appetite, Energy Intake, Butyrylcholinesterase Activity and Gut Peptides in Men With Variants of the Obesity-linked FTO rs9939609 Polymorphism
Brief Title: Effect of Exercise on Appetite, Gut Peptides and Butyrylcholinesterase Activity in Variants of the FTO Gene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: University College, London (Other); Rosetrees Trust (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Professor David Stensel, Professor of Exercise Metabolism, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: R14-P143
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Appetitive Behavior
MeSH Terms: conditions — Appetitive Behavior | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Experimental): Experimental day where participants rest.
  Interventions: Other: Control
- Exercise (Experimental): Experimental day where participants complete a run.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Control — Participants complete a resting control condition instead of a run.
  Arms: Control
Other: Exercise — Participants complete a 60 minute run at 70% of their maximal oxygen uptake
  Arms: Exercise

SUMMARY:
Using a database of individuals with FTO genetic data, the study aims to assess the appetite, energy intake, butyrylcholinesterase, gut hormone responses to a bout of moderate- to high intensity exercise in individuals with genetic variations in the FTO gene.

DETAILED DESCRIPTION:
The fat mass and obesity-associated gene (FTO) rs9939609 A allele is related to obesity, greater food intake and impaired postprandial reduction of ghrelin. Exercise acutely suppresses levels of ghrelin and appetite, yet whether the response differs in people with or without the rs9939609 A allele is unknown. This study assessed the effect of exercise on appetite, appetite-regulatory hormones and energy intake in variants of the FTO rs9939609 polymorphism.

Cohort

The investigators initially recruited 202 subjects to a database and measured FTO rs9939609 genotype. From these subjects, 12 individuals homozygous for the 'obesity-risk' rs9939609 A allele and 12 homozygous for the T allele were recruited.

A sample size of 24 was chosen based on previous data which suggested that a 34 pg/ml reduction in circulating acylated ghrelin during exercise could be detected with > 80% power with a two-tailed t-test whilst assuming a standard deviation of differences of 54 pg/ml.

Familiarisation trial

First, participants will arrive for a familiarisation trial. Participants will have been fasted for ~2-3 hours beforehand. Participant's height, weight and skinfold measures will be taken. Furthermore, a food preferences questionnaire will be completed to ensure the acceptability of food items provided during the study.

Participants will complete a sub-maximal fitness test, which will last for 16 minutes, and will comprise of four, four minute stages. Initial treadmill speed will be set according to fitness and will be increased every four minutes by 0.5-1.5 km/h. Prior to this test, participants will be fitted with a cannula into an antecubital vein and a blood sample will be withdrawn after the test. This will familiarise participants with the procedure and reduce any stress related to the novelty of the first visit.

Next, a maximal fitness test will be conducted to measure maximal oxygen uptake. This will consist of an incremental protocol where the treadmill gradient will begin at 3.5% and will be increased by 2.5% every 3 minutes. The speed of treadmill will remain constant, and will be determined based on fitness levels. Though the duration of the test is typically 9-15 minutes, it will last until the participant reaches volitional exhaustion.

After the fitness test and adequate recovery time, participants will be presented with a buffet-style meal and instructed to eat until comfortably full and satisfied. To finish, participants will be given a calibrated set of weighing scales and instructions to standardize their food intake before each main trial.

Main trials

Each participant will complete two main trials separated by 7 days: an exercise trial and control trial. In the 24 hours before a main trial, participants will follow a set of standardization procedures. Participants will record all foods consumed and the timings of meals before the first trial. This will be subsequently replicated in the 24 hours prior to the second main trial. Moreover, participants will visit the lab to be provided with a meal and will be instructed to prepare and consume between 19:00-20:00 the night before each main trial. Participants will also be instructed to refrain from strenuous physical activity and alcohol consumption during this period.

Participants will report to the lab on the morning of each trial at 08:00 following an overnight fast. Participants will be instructed to walk slowly to the lab in the morning of each trial.

At 08:30, a cannula will be inserted into an antecubital vein followed by 60 minutes of rest. On the exercise trial, from 09:30 to 10:30, participants will run at a continuous pace that corresponds to 70% of the participant's maximal oxygen uptake. Participants will rest on the bed during this same period of the control trial. Participants will rest and will be provided with a selection of movies to watch for the rest of the trial.

There will be two meals provided to the participants: a standardised meal and an ad libitum buffet style meal. The standardised meal will be a fixed breakfast meal that participants will be provided at 10:50, and will be instructed to consume within 20 minutes. The ad libitum buffet style meal will be given at 15:50 and will consist of an array of foods with differing energy and macronutrient compositions. Participants will be presented with the buffet foods for 30 minutes and will be instructed to eat until comfortably full and satisfied.

Statistical procedures

Linear mixed model, with factors being trial (exercise or control), genotype (AA or TT) and time will be performed on all time-course measures. Area under the curve will be calculated using the trapezoidal rule for outcome measures taken periodically throughout the day. Linear mixed models will also be used for trial and genotype comparisons of area under the curve values and measures not taken throughout the day. At points of interest, where significant main and interaction effects occur, post-hoc analysis was conducted using Holm-Bonferroni adjusted t-tests. Statistical significance was accepted as P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* non-smoker, not currently dieting, weight stable for >3 months (self-reported), no personal history of cardiovascular disease, metabolic disease or dyslipidaemia, European ancestry, no psychiatric or medical condition

Exclusion Criteria:

* food allergies, dislike or intolerance of study foods and drinks, irregular eating patterns, use of medication that could influence hormone concentrations

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Plasma acylated ghrelin concentrations (N=24) | 24 hours
  Measured using ELISA from venous blood samples
Plasma desacyl ghrelin concentrations (N=24) | 24 hours
  Measured using ELISA from venous blood samples
Subjective appetite (N=24) | 24 hours
  Measured using visual analogue scales
Ad-libitum energy intake (N=24) | 24 hours
  Measured at laboratory-based meals
Plasma butyrylcholinesterase activity (N=24) | First hour of main trial (three samples).
  Measured using Ellman's reagent protocol

SECONDARY OUTCOMES:
Plasma total glucagon-like peptide 1 concentrations (N=24) | 24 hours
  Measured using ELISA from venous blood samples
Plasma total peptide yy concentrations (N=24) | 24 hours
  Measured using ELISA from venous blood samples
Plasma leptin concentrations (N=24) | Baseline (fasting) sample
  Measured using ELISA from venous blood samples

CONTACTS AND LOCATIONS:
Overall Officials: David J Stensel, PhD, Principal Investigator — Loughborough University
Locations (1):
- Loughborough University, Loughborough, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frayling TM, Timpson NJ, Weedon MN, Zeggini E, Freathy RM, Lindgren CM, Perry JR, Elliott KS, Lango H, Rayner NW, Shields B, Harries LW, Barrett JC, Ellard S, Groves CJ, Knight B, Patch AM, Ness AR, Ebrahim S, Lawlor DA, Ring SM, Ben-Shlomo Y, Jarvelin MR, Sovio U, Bennett AJ, Melzer D, Ferrucci L, Loos RJ, Barroso I, Wareham NJ, Karpe F, Owen KR, Cardon LR, Walker M, Hitman GA, Palmer CN, Doney AS, Morris AD, Smith GD, Hattersley AT, McCarthy MI. A common variant in the FTO gene is associated with body mass index and predisposes to childhood and adult obesity. Science. 2007 May 11;316(5826):889-94. doi: 10.1126/science.1141634. Epub 2007 Apr 12. PMID 17434869
- [Background] Speakman JR, Rance KA, Johnstone AM. Polymorphisms of the FTO gene are associated with variation in energy intake, but not energy expenditure. Obesity (Silver Spring). 2008 Aug;16(8):1961-5. doi: 10.1038/oby.2008.318. Epub 2008 Jun 12. PMID 18551109
- [Background] Karra E, O'Daly OG, Choudhury AI, Yousseif A, Millership S, Neary MT, Scott WR, Chandarana K, Manning S, Hess ME, Iwakura H, Akamizu T, Millet Q, Gelegen C, Drew ME, Rahman S, Emmanuel JJ, Williams SC, Ruther UU, Bruning JC, Withers DJ, Zelaya FO, Batterham RL. A link between FTO, ghrelin, and impaired brain food-cue responsivity. J Clin Invest. 2013 Aug;123(8):3539-51. doi: 10.1172/JCI44403. Epub 2013 Jul 15. PMID 23867619
- [Derived] Dorling JL, Clayton DJ, Jones J, Carter WG, Thackray AE, King JA, Pucci A, Batterham RL, Stensel DJ. A randomized crossover trial assessing the effects of acute exercise on appetite, circulating ghrelin concentrations, and butyrylcholinesterase activity in normal-weight males with variants of the obesity-linked FTO rs9939609 polymorphism. Am J Clin Nutr. 2019 Nov 1;110(5):1055-1066. doi: 10.1093/ajcn/nqz188. PMID 31504106